CLINICAL TRIAL: NCT02522273
Title: Evaluation of the 'SensPoint' Lactate Meter Validation of a Hand-Held Lactate Measuring System 'SensPoint' in the Estimation of Foetal Scalp Blood and Umbilical Cord Blood Lactate
Brief Title: Evaluation of the 'SensPoint' Lactate Meter in the Estimation of Foetal Scalp Blood and Umbilical Cord Blood Lactate
Status: Withdrawn | Type: Observational
Sponsor: North Bristol NHS Trust (Other)
Collaborators: EKF Diagnostics (Unknown)
Responsible Party: Principal Investigator, Jo Crofts, Dr Joanna Crofts, North Bristol NHS Trust
Other Study IDs: 3493
Record Dates: First submitted 2015-08-10; First posted 2015-08-13 (Estimated); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Measurement of Fetal Blood Lactate
Keywords: Obstetric; Midwifery; Fetal blood sample; Lactate; Handheld meter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: EKF Diagnostics 'SensPoint' Lactate Meter

SUMMARY:
A cardiotocograph (CTG) can be used in labour to assess the heartbeat and well-being of a baby. An abnormal CTG may be a sign that a baby has low oxygen levels (hypoxia) and is becoming distressed.

In this situation a blood test can be taken from the scalp of the baby. A high lactate level in the blood indicates that urgent delivery is required to prevent long-term harm to the newborn.

SensPoint is a new medical device that measures lactate. It has several potential benefits over the current method of measuring lactate in that it is a portable hand-held device (allowing for use in the delivery room), requires a much smaller volume of blood and produces results more quickly than the current method of measuring lactate.

Before a new device is adopted into clinical practice, it is important that it is first confirmed that it is accurate and reliable for its intended use. This study will evaluate the ability of the SensPoint device to accurately and reliably detect lactate in fetal and umbilical cord blood by comparing its performance to the reference device currently in use.

DETAILED DESCRIPTION:
A cardiotocograph (CTG) can be used in labour to assess the heartbeat and well-being of a baby. An abnormal CTG may be a sign that a baby has low oxygen levels (hypoxia) and is becoming distressed.

In this situation a blood test can be taken from the scalp of the baby. A high lactate level or high acidity (low pH) in the blood indicates that urgent delivery is required to prevent long-term harm to the newborn.

Obtaining scalp blood can be difficult, time consuming and has a high failure rate. In the UK the majority of maternity units (including at North Bristol NHS Trust) will use a blood gas analyser to measure lactate. These are generally large, non-transportable devices located in or nearby the maternity unit. The blood gas analyser requires relatively large drops of baby's blood and due to it's fixed location, requires the midwife to leave the delivery room to process. Samples that are too small or contain air bubbles and blood clots will be rejected and need repeating. The process can take up to twenty minutes to complete.

After delivery blood from the umbilical cord is routinely obtained in high-risk deliveries for the measurement of pH and lactate. This establishes the wellbeing of the baby at the time of birth and can guide on-going treatment. Lactate in these samples is also measured using the blood gas analyser.

SensPoint is a new medical device that measures lactate. It has several potential benefits over the current method of measuring lactate in that it is a portable hand-held device (allowing for use in the delivery room), requires a much smaller volume of blood and produces results more quickly than the current method of measuring lactate.

Before a new device is adopted into clinical practice, it is important that it is first confirmed that it is accurate and reliable for its intended use. The researchers propose a study that will evaluate the ability of the SensPoint device to accurately and reliably detect lactate in both the laboratory and clinical setting by comparing its performance to the reference device currently in use.

The study will be divided into three parts:

1. Comparison of the SensPoint device and the reference device in laboratory prepared samples.
2. Comparison of the SensPoint device and the reference device using small volumes of leftover blood from umbilical cord blood testing obtained during routine care.
3. Comparison of the SensPoint device and the reference device using small volumes of leftover blood from foetal scalp sampling obtained during routine care.

All foetal blood samples utilised in this study are surplus to clinical requirements and would otherwise be discarded. Retrospective consent will be obtained.

For the purposes of ensuring validity, reliability and repeatability of the device the researchers will test 90 laboratory standard samples, 90 arterial and venous cord blood samples and 90 foetal scalp capillary blood samples.

This study will enable the research team to design a larger study directly comparing the two methods of measuring lactate, assessing factors such as speed and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* women who have a fetal blood sample or umbilical cord blood sampling as part of their care during childbirth

Exclusion Criteria:

* women in Prison

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women who have a fetal blood sample or umbilical cord blood sample taken for the measurement of lactate as part of their care during childbirth.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Comparison of lactate level in blood obtained from the fetal scalp measured using a Senspoint handheld lactate meter and the current gold standard. | Within 5 minutes of obtaining blood sample
  Foetal blood sampling will be undertaken as clinically indicated by National Intrapartum Guidance and serum lactate will be measured in the usual manner using the current gold standard.
  Once the serum lactate has been measured using the current gold standard (and the sample are no longer clinically useful and would normally be discarded) any blood remaining in the capillary tube will be handed to the research team. A member of the research team will then process the sample using the new Senspoint device.
  Lactate readings from (i) the reference machine and (ii) the Senspoint device will be compared using a Bland-Altman plot, a difference plot used in analytical chemistry and biostatistics to analyze the agreement between two different assays.
Comparison of lactate level in blood obtained from the umbilical artery measured using a Senspoint handheld lactate meter and the current gold standard. | Within 5 minutes of obtaining blood sample
  Blood from the umbilical artery will be sampled as clinically indicated by National Intrapartum Guidance and serum lactate will be measured in the usual manner using the current gold standard.
  Once the serum lactate has been measured using the current gold standard (and the sample are no longer clinically useful and would normally be discarded) any blood remaining in the syringe will be handed to the research team. A member of the research team will then process the sample using the new Senspoint device.
  Lactate readings from (i) the reference machine and (ii) the Senspoint device will be compared using a Bland-Altman plot, a difference plot used in analytical chemistry and biostatistics to analyze the agreement between two different assays.
Comparison of lactate level in blood obtained from the umbilical vein measured using a Senspoint handheld lactate meter and the current gold standard. | Within 5 minutes of obtaining blood sample
  Blood from the umbilical vein will be sampled as clinically indicated by National Intrapartum Guidance and serum lactate will be measured in the usual manner using the current gold standard.
  Once the serum lactate has been measured using the current gold standard (and the sample are no longer clinically useful and would normally be discarded) any blood remaining in the syringe will be handed to the research team. A member of the research team will then process the sample using the new Senspoint device.
  Lactate readings from (i) the reference machine and (ii) the Senspoint device will be compared using a Bland-Altman plot, a difference plot used in analytical chemistry and biostatistics to analyze the agreement between two different assays.

CONTACTS AND LOCATIONS:
Locations (1):
- North Bristol NHS Trust, Bristol, United Kingdom